CLINICAL TRIAL: NCT05617183
Title: A Phase 1, Randomized, Open-label, Two-arm, Parallel Group, Single-dose Study to Compare the Pharmacokinetics and Safety of the Auto-injector and Pre-filled Syringe of CT-P47 in Healthy Subjects
Brief Title: Compare the Auto-injector and Pre-filled Syringe of CT-P47 in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CT-P47 1.3
Record Dates: First submitted 2022-10-25; First posted 2022-11-15 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CT-P47 Auto-injector (Experimental): CT-P47, 162 mg in 0.9 mL, a single subcutaneous (SC) injection via auto-injector (AI)
  Interventions: Biological: CT-P47
- CT-P47 Pre-filled Syringe (Active Comparator): CT-P47, 162 mg in 0.9 mL, a single subcutaneous (SC) injection via pre-filled syringe (PFS)
  Interventions: Biological: CT-P47

INTERVENTIONS:
Biological: CT-P47 — CT-P47, 162 mg in 0.9 mL, a single subcutaneous (SC) injection via auto-injector (AI)
  Arms: CT-P47 Auto-injector
Biological: CT-P47 — CT-P47, 162 mg in 0.9 mL, a single subcutaneous (SC) injection via pre-filled syringe (PFS)
  Arms: CT-P47 Pre-filled Syringe

SUMMARY:
This is a phase 1 study to compare the Pharmacokinetics and Safety of the Auto-injector and Pre-filled syringe of CT-P47 in Healthy Subjects.

DETAILED DESCRIPTION:
CT-P47, containing the active ingredient tocilizumab, is a recombinant humanized monoclonal antibody that is being developed as a similar biological medicinal product to RoActemra/Actemra. The purpose of this study is to demonstrate the pharmacokinetics and safety of the Auto-injector and Pre-filled syringe of CT-P47 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects between the ages of 19 to 55 years, both inclusive.
2. Subject with a body weight of ≥60 and ≤100 kg for male and ≥50 and ≤100 kg for female and a BMI between 18.5 and 28.0 kg/m2 (both inclusive) when rounded to the nearest tenth.

Exclusion Criteria:

1. A medical history and/or condition that is considered significant
2. Clinically significant allergic reactions, hypersensitivity
3. History or current infection of hepatitis B virus, hepatitis C virus, human immunodeficiency virus, or syphilis
4. Active or latent Tuberculosis
5. History of malignancy
6. Previous exposure to tocilizumab or any drug that targets IL-6

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 268 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
PK similarity demonstration by AUC | Day 43
  Demonstrate PK similarity in terms of area under the concentration-time curve (AUC) from time zero to infinity (AUC0-inf) of CT-P47 SC administration via AI versus PFS in healthy subjects up to Day 43. The similarity of PK between CT-P47 AI vs CT-P47 PFS will be concluded if the 90% Cls for the ratios of geometric means of the comparison are entirely contained within the equivalence margin of 80% to 125% for AUC0-inf.
PK similarity demonstration by Cmax | Day 43
  Demonstrate PK similarity in terms of maximum serum concentration (Cmax) of CT-P47 SC administration via AI versus PFS in healthy subjects up to Day 43. The similarity of PK between CT-P47 AI vs CT-P47 PFS will be concluded if the 90% Cls for the ratios of geometric means of the comparison are entirely contained within the equivalence margin of 80% to 125% for Cmax.

SECONDARY OUTCOMES:
Additional PK evaluation | Day 43
  Evaluate additional PK in terms of AUC from time zero to the last quantifiable concentration (AUC0-last).
Safety evaluation by TEAEs | Day 43
  Evaluate safety in terms of treatment-emergent adverse events (TEAEs) of CT-P47.

CONTACTS AND LOCATIONS:
Overall Officials: KyungSang Yu, Principal Investigator — Seoul National University College of Medicine and Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yu KS, Ryu H, Shin D, Park M, Hwang J, Moon SJ, Kim MG, Keystone E, Smolen JS, Kim S, Bae Y, Jeon D, Jang J, Yang G, Bae J, Lee J, Burmester GR. Pharmacokinetics and safety of candidate tocilizumab biosimilar CT-P47 administered by auto-injector or pre-filled syringe: a randomized, open-label, single-dose phase I study. Expert Opin Biol Ther. 2024 Jul;24(7):681-689. doi: 10.1080/14712598.2024.2321360. Epub 2024 Jun 21. PMID 38905143